CLINICAL TRIAL: NCT05627453
Title: Helping Older People Recover Walking Abilities Through Arm-in-armg Gait Training: a Randomized Controlled Trial
Brief Title: Arm-in-Arm Gait Training Trial
Acronym: AAGaTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philippe Terrier (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Philippe Terrier, Assistant professor, Haute Ecole ARC Sante
Organization: Haute Ecole ARC Sante (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-01452
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Healthy Aging
Keywords: fall risk; gait disorder; physical activity; complexity matching
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Intervention Model Description: The AAGaTT study, is a monocentric, two-arm, open-label, randomized controlled trial. The superiority of arm-in-arm synchronized gait training will be assessed versus standard walking (i.e., walking side-by-side without gait synchronization).
Masking Description: Blinding is not possible due to the nature of the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal gait training (Active Comparator): The gait training session will consist in 30 min walking side-by-side. If any, the session will take place along an indoor circuit to avoid unfavorable weather conditions. The participants will walk side by side without contact and without instructions about gait synchronisation. They will have to agree on a comfortable pace for the older participant.
  The gait training session will be repeated three times a week for four weeks. The last session of each week will also include an assessement of gait quality.
  Interventions: Other: Normal gait training
- Arm-in-arm gait training (Experimental): The gait training session will consist in 30 min walking side-by-side. If any, the session will take place along an indoor circuit to avoid unfavorable weather conditions. The participants will be asked to walk arm-in-arm while synchronizing their steps. They will have to agree on a comfortable pace for the older participant.
  The gait training session will be repeated three times a week for four weeks. The last session of each week will also include an assessement of gait quality.
  Interventions: Other: Arm-in-arm gait training

INTERVENTIONS:
Other: Arm-in-arm gait training — An older adult walk side-by-side, arm-in-arm with a younger adult while synchronizing steps.
  Arms: Arm-in-arm gait training
Other: Normal gait training — An older adult walk side-by-side, without contact, with a younger adult without step synchronization.
  Arms: Normal gait training

SUMMARY:
The AAGaTT study, is a monocentric, two-arm, open-label, randomized controlled trial. The objective is to assess the efficacy of an arm-in-arm walking program for older people at risk of falling. Gait training imply that the older participants must walk while synchronizing steps with a younger partner.

DETAILED DESCRIPTION:
A high level of physical activity is the cornerstone of healthy aging. Falls are a major issue in elderly population, and exercising can mitigate their occurrence. However, the type of exercise-and the optimal way to deliver it-that maximises efficacy is still unknown. The ideal-most efficient-exercise intervention should have the following characteristics: it should have a specific effect on fall risk mitigation, it should be of sufficient intensity to improve cardiovascular fitness and muscle strength, it should be safe, it should not induce high costs, and it should be sufficiently enjoyable and motivational to induce a high adherence and compliance. The present trial aims at testing an innovative exercise intervention that may exhibit all these advantages.

The intervention will consist in four weeks of 30min arm-in-arm synchronized gait training three times a week. Convincing evidence from the literature supports the use of rhythmic externals cues, either auditory or visual, to improve the efficacy of gait training for fall risk reduction in seniors. Synchronizing gait with a younger partner may bring further benefits.

We will focus on clinically relevant outcomes to highlight potential benefits of the intervention in term of gait quality, balance, fall risk mitigation, physical activity level, mood, and well-being.

Gait quality will be assessed through two inertial sensors attached to the low back and foot. Six gait assessement sessions are planned: at baseline (before randomization), at the end of each training week, and at week 7 (follow-up). Participants will walk at their preferred speed over 200m.

We will also include functional tests and self-filled questionnaires to evaluate participant's abilities and mood.

Falls occuring within 18 months after inclusion will be tracked via an online questionnaire every three months.

We will assess the superiority of arm-in-arm gait training compared to standard walking (without gait synchronisation) via a randomized-controlled design. The perception of the intervention by elderly participants will be explored via a qualitative analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Older Participant

   * Older than 70 years old
   * Able to walk continuously during 15 minutes without walking aids.
   * Must have experienced a fall during the last year before the recruitment.
   * Health certificate that attests no contraindication to walking
   * No severe gait disorders from orthopedic or neurologic origins (such as lower-limb amputation or severe hemiparesis). Mild gait abnormalities (for example, mild limping due to knee arthritis, or slight gait asymmetry due to limited hemiparesis) will be tolerated.
2. Younger Participant

   * Older than 18 years old but younger than 40 years old.
   * No severe gait disorders from musculoskeletal or neurologic origin.

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc.;
* Inability or contraindications to undergo the investigated intervention.
* Vulnerable persons, in sense of swiss Human Research Act art. 21-24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Walking speed | Week 4
  Habitual (preferred) walking speed to cover 200m. Normal values for older men: 1.21m/s -1.32m/s), older women 1.07m/s -1.19m/s).

SECONDARY OUTCOMES:
Walking speed | Baseline
  Habitual (preferred) walking speed to cover 200m. Normal values for older men: 1.21m/s -1.32m/s), older women 1.07m/s -1.19m/s).
Walking speed | Week 1
  Habitual (preferred) walking speed to cover 200m. Normal values for older men: 1.21m/s -1.32m/s), older women 1.07m/s -1.19m/s).
Walking speed | Week 2
  Habitual (preferred) walking speed to cover 200m. Normal values for older men: 1.21m/s -1.32m/s), older women 1.07m/s -1.19m/s).
Walking speed | Week 3
  Habitual (preferred) walking speed to cover 200m. Normal values for older men: 1.21m/s -1.32m/s), older women 1.07m/s -1.19m/s).
Walking speed | Week 7 (follow-up)
  Habitual (preferred) walking speed to cover 200m. Normal values for older men: 1.21m/s -1.32m/s), older women 1.07m/s -1.19m/s).
Average step frequency | Baseline
  Average number of steps per second while walking at habitual (preferred) speed over 200m.
Step frequency | Week 1
  Average number of steps per second while walking at habitual (preferred) speed over 200m.
Step frequency | Week 2
  Average number of steps per second while walking at habitual (preferred) speed over 200m.
Step frequency | Week 3
  Average number of steps per second while walking at habitual (preferred) speed over 200m.
Step frequency | Week 4
  Average number of steps per second while walking at habitual (preferred) speed over 200m.
Step frequency | Week 7 (follow-up)
  Average number of steps per second while walking at habitual (preferred) speed over 200m.
Step length | Baseline
  Average step length while walking at habitual (preferred) speed over 200m.
Step length | Week 1
  Average step length while walking at habitual (preferred) speed over 200m.
Step length | Week 2
  Average step length while walking at habitual (preferred) speed over 200m.
Step length | Week 3
  Average step length while walking at habitual (preferred) speed over 200m.
Step length | Week 4
  Average step length while walking at habitual (preferred) speed over 200m.
Step length | Week 7 (follow-up)
  Average step length while walking at habitual (preferred) speed over 200m.
Step symmetry | Baseline
  Left / right symmetry of the gait assessed via the autocorrelation method. A high value shows a symmetric gait.
Step symmetry | Week 1
  Left / right symmetry of the gait assessed via the autocorrelation method. A high value shows a symmetric gait.
Step symmetry | Week 2
  Left / right symmetry of the gait assessed via the autocorrelation method. A high value shows a symmetric gait.
Step symmetry | Week 3
  Left / right symmetry of the gait assessed via the autocorrelation method. A high value shows a symmetric gait.
Step symmetry | Week 4
  Left / right symmetry of the gait assessed via the autocorrelation method. A high value shows a symmetric gait.
Step symmetry | Week 7 (follow-up)
  Left / right symmetry of the gait assessed via the autocorrelation method. A high value shows a symmetric gait.
Stride regularity | Baseline
  Left / right symmetry of the gait assessed via the autocorrelation method. A high value shows a symmetric gait.
Stride regularity | Week 1
  Left / right symmetry of the gait assessed via the autocorrelation method. A high value shows a symmetric gait.
Stride regularity | Week 2
  Regularity of the gait assessed via the autocorrelation method. A high value shows a less variable gait.
Stride regularity | Week 3
  Regularity of the gait assessed via the autocorrelation method. A high value shows a less variable gait.
Stride regularity | Week 4
  Regularity of the gait assessed via the autocorrelation method. A high value shows a less variable gait.
Stride regularity | Week 7 (follow-up)
  Regularity of the gait assessed via the autocorrelation method. A high value shows a less variable gait.
Gait Stability | Baseline
  short-term Local dynamic stability (maximal Lyapunov exponent). A low value shows a more stable gait and a lower risk of fall.
Gait Stability | Week 1
  short-term Local dynamic stability (maximal Lyapunov exponent). A low value shows a more stable gait and a lower risk of fall.
Gait Stability | Week 2
  short-term Local dynamic stability (maximal Lyapunov exponent). A low value shows a more stable gait and a lower risk of fall.
Gait Stability | Week 3
  short-term Local dynamic stability (maximal Lyapunov exponent). A low value shows a more stable gait and a lower risk of fall.
Gait Stability | Week 4
  short-term Local dynamic stability (maximal Lyapunov exponent). A low value shows a more stable gait and a lower risk of fall.
Gait Stability | Week 7 (follow-up)
  short-term Local dynamic stability (maximal Lyapunov exponent). A low value shows a more stable gait and a lower risk of fall.
Gait attentional demand | Baseline
  Attractor complexity index. A high value indicates that less attention is dedicated to control gait (automated gait).
Gait attentional demand | Week 1
  Attractor complexity index. A high value indicates that less attention is dedicated to control gait (automated gait).
Gait attentional demand | Week 2
  Attractor complexity index. A high value indicates that less attention is dedicated to control gait (automated gait).
Gait attentional demand | Week 3
  Attractor complexity index. A high value indicates that less attention is dedicated to control gait (automated gait).
Gait attentional demand | Week 4
  Attractor complexity index. A high value indicates that less attention is dedicated to control gait (automated gait).
Gait attentional demand | Week 7 (follow-up)
  Attractor complexity index. A high value indicates that less attention is dedicated to control gait (automated gait).
Fractal index | Baseline
  Attentional demand measured via detrended fluctuation analysis (DFA). A high value indicates that less attention is dedicated to control gait (automated gait).
Fractal index | Week 1
  Attentional demand measured via detrended fluctuation analysis (DFA). A high value indicates that less attention is dedicated to control gait (automated gait).
Fractal index | Week 2
  Attentional demand measured via detrended fluctuation analysis (DFA).A high value indicates that less attention is dedicated to control gait (automated gait).
Fractal index | Week 3
  Attentional demand measured via detrended fluctuation analysis (DFA).A high value indicates that less attention is dedicated to control gait (automated gait).
Fractal index | Week 4
  Attentional demand measured via detrended fluctuation analysis (DFA).A high value indicates that less attention is dedicated to control gait (automated gait).
Fractal index | Week 7 (follow-up)
  Attentional demand measured via detrended fluctuation analysis (DFA).A high value indicates that less attention is dedicated to control gait (automated gait).
Stride time variability | Baseline
  Variability of stride (gait cycle) duration over 200m walking. A high value shows a high stride-to-stride variability.
Stride time variability | Week 1
  Variability of stride (gait cycle) duration over 200m walking. A high value shows a high stride-to-stride variability.
Stride time variability | Week 2
  Variability of stride (gait cycle) duration over 200m walking. A high value shows a high stride-to-stride variability.
Stride time variability | Week 3
  Variability of stride (gait cycle) duration over 200m walking. A high value shows a high stride-to-stride variability.
Stride time variability | Week 4
  Variability of stride (gait cycle) duration over 200m walking. A high value shows a high stride-to-stride variability.
Stride time variability | Week 7 (follow-up)
  Variability of stride (gait cycle) duration over 200m walking. A high value shows a high stride-to-stride variability.
Time to perform Timed up-and-go (TUG) test. | Baseline
  The Timed Up and Go (TUG) test is a clinical test used to assess balance and walking ability in older populations. The test measures the time a participant take to get up from an armed chair, walk three meters to a line drawn on the floor, turn around and sit back down in the same chair. The time is measured in seconds.
  The results can be interpreted the following way:
  * ≤ 10 seconds = normal, good general health
  * ≤ 20 seconds = good mobility, can go out alone, mobile without a gait aid
  * > 30 seconds = difficulties, cannot go outside alone, requires a gait aid
Time to perform Timed up-and-go (TUG) test. | Week 1
  The Timed Up and Go (TUG) test is a clinical test used to assess balance and walking ability in older populations. The test measures the time a participant take to get up from an armed chair, walk three meters to a line drawn on the floor, turn around and sit back down in the same chair. The time is measured in seconds.
  The results can be interpreted the following way:
  * ≤ 10 seconds = normal, good general health
  * ≤ 20 seconds = good mobility, can go out alone, mobile without a gait aid
  * > 30 seconds = difficulties, cannot go outside alone, requires a gait aid
Time to perform Timed up-and-go (TUG) test. | Week 2
  The Timed Up and Go (TUG) test is a clinical test used to assess balance and walking ability in older populations. The test measures the time a participant take to get up from an armed chair, walk three meters to a line drawn on the floor, turn around and sit back down in the same chair. The time is measured in seconds.
  The results can be interpreted the following way:
  * ≤ 10 seconds = normal, good general health
  * ≤ 20 seconds = good mobility, can go out alone, mobile without a gait aid
  * > 30 seconds = difficulties, cannot go outside alone, requires a gait aid
Time to perform Timed up-and-go (TUG) test. | Week 3
  The Timed Up and Go (TUG) test is a clinical test used to assess balance and walking ability in older populations. The test measures the time a participant take to get up from an armed chair, walk three meters to a line drawn on the floor, turn around and sit back down in the same chair. The time is measured in seconds.
  The results can be interpreted the following way:
  * ≤ 10 seconds = normal, good general health
  * ≤ 20 seconds = good mobility, can go out alone, mobile without a gait aid
  * > 30 seconds = difficulties, cannot go outside alone, requires a gait aid
Time to perform the Timed up-and-go (TUG) test. | Week 4
  The Timed Up and Go (TUG) test is a clinical test used to assess balance and walking ability in older populations. The test measures the time a participant take to get up from an armed chair, walk three meters to a line drawn on the floor, turn around and sit back down in the same chair. The time is measured in seconds.
  The results can be interpreted the following way:
  * ≤ 10 seconds = normal, good general health
  * ≤ 20 seconds = good mobility, can go out alone, mobile without a gait aid
  * > 30 seconds = difficulties, cannot go outside alone, requires a gait aid
Time to perform the Timed up-and-go (TUG) test. | Week 7 (follow-up)
  The Timed Up and Go (TUG) test is a clinical test used to assess balance and walking ability in older populations. The test measures the time a participant take to get up from an armed chair, walk three meters to a line drawn on the floor, turn around and sit back down in the same chair. The time is measured in seconds.
  The results can be interpreted the following way:
  * ≤ 10 seconds = normal, good general health
  * ≤ 20 seconds = good mobility, can go out alone, mobile without a gait aid
  * > 30 seconds = difficulties, cannot go outside alone, requires a gait aid
Average time held on a leg obtained following the Unipedal stance test | Baseline
  The Unipedal stance test measure the ability to stand on one leg and maintain balance. The participants are asked to stand as long as possible on one leg. The exercise is repeated three times for each leg. The time is measure in seconds. The average of the scores is calculated.
  The mean time held for people aged 70-79 is 14.2 +/- 9.3 seconds.
Average time held on a leg obtained following the Unipedal stance test | Week 1
  The Unipedal stance test measure the ability to stand on one leg and maintain balance. The participants are asked to stand as long as possible on one leg. The exercise is repeated three times for each leg. The time is measure in seconds. The average of the scores is calculated.
  The mean time held for people aged 70-79 is 14.2 +/- 9.3 seconds.
Average time held on a leg obtained following the Unipedal stance test | Week 2
  The Unipedal stance test measure the ability to stand on one leg and maintain balance. The participants are asked to stand as long as possible on one leg. The exercise is repeated three times for each leg. The time is measure in seconds. The average of the scores is calculated.
  The mean time held for people aged 70-79 is 14.2 +/- 9.3 seconds.
Average time held on a leg obtained following the Unipedal stance test | Week 3
  The Unipedal stance test measure the ability to stand on one leg and maintain balance. The participants are asked to stand as long as possible on one leg. The exercise is repeated three times for each leg. The time is measure in seconds. The average of the scores is calculated.
  The mean time held for people aged 70-79 is 14.2 +/- 9.3 seconds.
Average time held on a leg obtained following the Unipedal stance test | Week 4
  The Unipedal stance test measure the ability to stand on one leg and maintain balance. The participants are asked to stand as long as possible on one leg. The exercise is repeated three times for each leg. The time is measure in seconds. The average of the scores is calculated.
  The mean time held for people aged 70-79 is 14.2 +/- 9.3 seconds.
Average time held on a leg obtained accordion to the Unipedal stance test | Week 7 (follow-up)
  The Unipedal stance test measure the ability to stand on one leg and maintain balance. The participants are asked to stand as long as possible on one leg. The exercise is repeated three times for each leg. The time is measure in seconds. The average of the scores is calculated.
  The mean time held for people aged 70-79 is 14.2 +/- 9.3 seconds.
Score at the Geriatric Depression Scale (GDS) | Baseline
  The Geriatric Depression Scale (GDS) is a self-rating scale designed for rating depression in older adults. The GDS questionnaire is composed of 15 questions. 10 of the questions indicate the presence of depression when answered positively, the 5 others indicate the presence of depression if answered negatively.
  * A score between 0 and 5 indicate a normal state.
  * A score between 5 and 11 indicate a mild to moderate depression.
  * A score between 11 and 15 indicate a severe depression.
Score at the Geriatric Depression Scale (GDS) | Week 4
  The Geriatric Depression Scale (GDS) is a self-rating scale designed for rating depression in older adults. The GDS questionnaire is composed of 15 questions. 10 of the questions indicate the presence of depression when answered positively, the 5 others indicate the presence of depression if answered negatively.
  * A score between 0 and 5 indicate a normal state.
  * A score between 5 and 11 indicate a mild to moderate depression.
  * A score between 11 and 15 indicate a severe depression.
Score at the Geriatric Depression Scale (GDS) | Week 7 (follow-up)
  The Geriatric Depression Scale (GDS) is a self-rating scale designed for rating depression in older adults. The GDS questionnaire is composed of 15 questions. 10 of the questions indicate the presence of depression when answered positively, the 5 others indicate the presence of depression if answered negatively.
  * A score between 0 and 5 indicate a normal state.
  * A score between 5 and 11 indicate a mild to moderate depression.
  * A score between 11 and 15 indicate a severe depression.
Score at the Falls Efficacy Scale International (FES-I) | Baseline
  The FES-I questionnaire measure the "concern about falling". The questionnaire is composed of 16 questions with 4 choices valued from 1 to 4: "not at all concerned" (1), "a little concerned" (2), "somewhat concerned" (3), and "very concerned" (4). The minimum score is 16 and the highest 64.
  * A score between 16 and 19 indicate a low concern about falling.
  * A score between 20 and 27 indicates a moderate concern about falling.
  * A score above 28 indicates a high concern about falling.
Score at the Falls Efficacy Scale International (FES-I) | Week 4
  The FES-I questionnaire measure the "concern about falling". The questionnaire is composed of 16 questions with 4 choices valued from 1 to 4: "not at all concerned" (1), "a little concerned" (2), "somewhat concerned" (3), and "very concerned" (4). The minimum score is 16 and the highest 64.
  * A score between 16 and 19 indicate a low concern about falling.
  * A score between 20 and 27 indicates a moderate concern about falling.
  * A score above 28 indicates a high concern about falling.
Score at the Falls Efficacy Scale International (FES-I) | Week 7 (follow-up)
  The FES-I questionnaire measure the "concern about falling". The questionnaire is composed of 16 questions with 4 choices valued from 1 to 4: "not at all concerned" (1), "a little concerned" (2), "somewhat concerned" (3), and "very concerned" (4). The minimum score is 16 and the highest 64.
  * A score between 16 and 19 indicate a low concern about falling.
  * A score between 20 and 27 indicates a moderate concern about falling.
  * A score above 28 indicates a high concern about falling.
Level of physical activity over the last seven days | Baseline
  The "Questionnaire d'activité physique pour les personnes âgées (QAPPA)" evaluates the level of physical activity (LoPA) over the last 7days. Moderate (M) and Vigorous (V) physical activity (PA) are distinguished. The time spent per week (minutes) is multiplied by 8 for V activities and by 4 for the M activities and indicate the level of MET-min/week (Metabolic Equivalent of Task).
  Moderate LoPA:
  1. 150 minutes of PA (M, V or both) spread over at least 3 days of the last 7 days.
  2. 800 MET-min/week of PA (M, V, or both) spread over 2 days of the last 7 days.
  3. At least 20 minutes of V PA spread over 3 days of the last 7 days.
  High LoPA:
  1. At least 1500 MET-min/week of V PA spread over 3 days of the last 7 days
  2. At least 3000 MET-min/week of M, V, or both, PA spread over 3 days of the last 7 days.
  Low LoPA: cases that do not meet the classification for moderate or high level of activity.
Level of physical activity over the last seven days | Week 4
  The "Questionnaire d'activité physique pour les personnes âgées (QAPPA)" evaluates the level of physical activity (LoPA) over the last 7days. Moderate (M) and Vigorous (V) physical activity (PA) are distinguished. The time spent per week (minutes) is multiplied by 8 for V activities and by 4 for the M activities and indicate the level of MET-min/week (Metabolic Equivalent of Task).
  Moderate LoPA:
  1. 150 minutes of PA (M, V or both) spread over at least 3 days of the last 7 days.
  2. 800 MET-min/week of PA (M, V, or both) spread over 2 days of the last 7 days.
  3. At least 20 minutes of V PA spread over 3 days of the last 7 days.
  High LoPA:
  1. At least 1500 MET-min/week of V PA spread over 3 days of the last 7 days
  2. At least 3000 MET-min/week of M, V, or both, PA spread over 3 days of the last 7 days.
  Low LoPA: cases that do not meet the classification for moderate or high level of activity.
Level of physical activity over the last seven days | Week 7 (follow-up)
  The "Questionnaire d'activité physique pour les personnes âgées (QAPPA)" evaluates the level of physical activity (LoPA) over the last 7days. Moderate (M) and Vigorous (V) physical activity (PA) are distinguished. The time spent per week (minutes) is multiplied by 8 for V activities and by 4 for the M activities and indicate the level of MET-min/week (Metabolic Equivalent of Task).
  Moderate LoPA:
  1. 150 minutes of PA (M, V or both) spread over at least 3 days of the last 7 days.
  2. 800 MET-min/week of PA (M, V, or both) spread over 2 days of the last 7 days.
  3. At least 20 minutes of V PA spread over 3 days of the last 7 days.
  High LoPA:
  1. At least 1500 MET-min/week of V PA spread over 3 days of the last 7 days
  2. At least 3000 MET-min/week of M, V, or both, PA spread over 3 days of the last 7 days.
  Low LoPA: cases that do not meet the classification for moderate or high level of activity.
Measure of the quality of life and well-being | Baseline
  The Investigating Choice Experiments for the Preferences of Older People (ICEPOP) CAPability (ICECAP-O) is a capability-based measure of the general quality of life of older people (≥ 65 years old). The ICECAP-O measures 5 attributes,each attribute has 4 level of answers. The 20 ICECAP-O attribute levels are estimated independently of one another such as the lowest level of capability (no capability on all attributes) was given a total value of 0 and the highest level of capability (full capability on all attributes) was given a total value of 1. The ICEPCAP-O range on a scale from 0 to 1.
Measure of the quality of life and well-being | Week 4
  The Investigating Choice Experiments for the Preferences of Older People (ICEPOP) CAPability (ICECAP-O) is a capability-based measure of the general quality of life of older people (≥ 65 years old). The ICECAP-O measures 5 attributes,each attribute has 4 level of answers. The 20 ICECAP-O attribute levels are estimated independently of one another such as the lowest level of capability (no capability on all attributes) was given a total value of 0 and the highest level of capability (full capability on all attributes) was given a total value of 1. The ICEPCAP-O range on a scale from 0 to 1.
Number of falls over the past year | Baseline
  The number of falls over the past year will be use to determine the retrospective fall rate.
Number of falls over three months | Between 0 and 3 months after the end of the training program (week 4).
  The number of falls over three month will be used to determine the prospective fall rate. The measure will be taken every three month until 18 moths after the beginning of the training program or in the case the participants felt two times between the measure and the end of the training program.
Number of falls over three month | Between 3 and 6 months after the end of the training program (week 4).
  The number of falls over three month will be used to determine the prospective fall rate. The measure will be taken every three month until 18 moths after the beginning of the training program or in the case the participants felt two times between the measure and the end of the training program.
Number of falls over three months | Between 6 and 9 months after the end of the training program (week 4).
  The number of falls over three month will be used to determine the prospective fall rate. The measure will be taken every three month until 18 moths after the beginning of the training program or in the case the participants felt two times between the measure and the end of the training program.
Number of falls over three months | Between 9 and 12 months after the end of the training program (week 4).
  The number of falls over three month will be used to determine the prospective fall rate. The measure will be taken every three month until 18 moths after the beginning of the training program or in the case the participants felt two times between the measure and the end of the training program.
Number of falls over three months | Between 12 and 15 months after the end of the training program (week 4).
  The number of falls over three month will be used to determine the prospective fall rate. The measure will be taken every three month until 18 moths after the beginning of the training program or in the case the participants felt two times between the measure and the end of the training program.
Number of falls over three months | Between 12 and 18 months after the end of the training program (week 4).
  The number of falls over three month will be used to determine the prospective fall rate. The measure will be taken every three month until 18 moths after the beginning of the training program or in the case the participants felt two times between the measure and the end of the training program.
Perception of the training program | Week 4
  Narrative feedback after transcription of semi-structured interviews. Quotes will be chosen to demonstrate themes which were common, or which represented a summary of a topic.
Number of participants withdrawing from the study | Week 7 (follow-up)
  The number of participants withdrawing from the study will be used to measure the adherence to the training program.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Terrier, PhD, Principal Investigator — Haute-Ecole Arc
Locations (1):
- Haute-Ecole Arc Santé, Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the final dataset will be anonymized. The anonymization process will constitute in the replacement of the participant unique ID (identification) by a random number.
  The acceleration data will be publicly shared on an online digital data repository (Zenodo: https://zenodo.org/).
  The shared data will not contain identification information; that is, shared personal data will be restricted to sex, body mass, body height, and age at time of the experiment (rounded year). Only the overall scores of questionnaires will be shared. Regarding the results of the qualitative study, only the anonymized transcripts will be shared. The audio files will be erased after the end of the study.
  The study protocol will be published in an open-access journal.
Supporting Information: Study Protocol
Time Frame: Study protocol will be published within 6 months after first recruitment. Anonymized dataset and acceleration data will be uploaded in parallel of result publications, within one year after the end of the study
Access Criteria: Study shared data will be publicly available on an open-access website following the FAIR (Findability, Accessibility, Interoperability, and Reuse) principles (zenodo.org).

REFERENCES:
- [Background] Ghai S, Ghai I, Effenberg AO. Effect of Rhythmic Auditory Cueing on Aging Gait: A Systematic Review and Meta-Analysis. Aging Dis. 2018 Oct 1;9(5):901-923. doi: 10.14336/AD.2017.1031. eCollection 2018 Oct. PMID 30271666
- [Background] Van Abbema R, De Greef M, Craje C, Krijnen W, Hobbelen H, Van Der Schans C. What type, or combination of exercise can improve preferred gait speed in older adults? A meta-analysis. BMC Geriatr. 2015 Jul 1;15:72. doi: 10.1186/s12877-015-0061-9. PMID 26126532
- [Background] Sherrington C, Fairhall NJ, Wallbank GK, Tiedemann A, Michaleff ZA, Howard K, Clemson L, Hopewell S, Lamb SE. Exercise for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD012424. doi: 10.1002/14651858.CD012424.pub2. PMID 30703272
- [Background] Almurad ZMH, Roume C, Blain H, Delignieres D. Complexity Matching: Restoring the Complexity of Locomotion in Older People Through Arm-in-Arm Walking. Front Physiol. 2018 Dec 4;9:1766. doi: 10.3389/fphys.2018.01766. eCollection 2018. PMID 30564149
- [Background] Terrier P, Le Carre J, Connaissa ML, Leger B, Luthi F. Monitoring of Gait Quality in Patients With Chronic Pain of Lower Limbs. IEEE Trans Neural Syst Rehabil Eng. 2017 Oct;25(10):1843-1852. doi: 10.1109/TNSRE.2017.2688485. Epub 2017 Mar 28. PMID 28368823
- [Background] Terrier P, Reynard F. Maximum Lyapunov exponent revisited: Long-term attractor divergence of gait dynamics is highly sensitive to the noise structure of stride intervals. Gait Posture. 2018 Oct;66:236-241. doi: 10.1016/j.gaitpost.2018.08.010. Epub 2018 Aug 14. PMID 30212783
- [Background] Bohannon RW, Williams Andrews A. Normal walking speed: a descriptive meta-analysis. Physiotherapy. 2011 Sep;97(3):182-9. doi: 10.1016/j.physio.2010.12.004. Epub 2011 May 11. PMID 21820535
- [Derived] Gigonzac M, Terrier P. Restoring walking ability in older adults with arm-in-arm gait training: study protocol for the AAGaTT randomized controlled trial. BMC Geriatr. 2023 Sep 6;23(1):542. doi: 10.1186/s12877-023-04255-9. PMID 37674129